CLINICAL TRIAL: NCT06767098
Title: The Effect of Mobile Holder in Treatment of Patients with Non-Specific Neck Pain.
Brief Title: Efficacy of New Ergonomic Device in Non-Specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, omnia mohamed, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005574
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Neck Pain
Keywords: neck pain; text neck; smartphone; ergonomics; posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditional therapeutic exercise for neck pain and smartphone holder (Experimental): Strech exercise for tight muscles as trapezius and levator scapulae. strengthening exercises for deep neck flexor and neck extensors. instructions to use a smartphone holder.
  Interventions: Other: theraputic exercises for neck muscles and smartphone holder
- traditional therapeutic exercise for neck pain (Active Comparator): Strech exercise for tight muscles as trapezius and levator scapulae. strengthening exercises for deep neck flexor and neck extensors.
  Interventions: Other: theraputic exercises for neck muscles

INTERVENTIONS:
Other: theraputic exercises for neck muscles and smartphone holder — strech and strength exercises for neck muscles. and using smartphone holder daily.
  Arms: traditional therapeutic exercise for neck pain and smartphone holder
Other: theraputic exercises for neck muscles — strech and strength exercises for neck muscles.
  Arms: traditional therapeutic exercise for neck pain

SUMMARY:
The goal of this clinical trial is to learn if smartphone holder works to treat neck pain in adults. It will also learn about the usability of smartphone holders. The main questions it aims to answer are:

* Does the smartphone holder decrease pain level and improve function in case of neck pain?
* How likely will the participants recommend the holder for their friends?

Researchers will compare adding the holder to the commonly used exercises for neck pain to a group which will receive the common exercise only. To see if the holder can modify neck pain.

Participants will:

* Do the exercise with or without using the holder
* Visit the clinic 3 times per week for a month for receiving exercise
* Keep a diary of their usage for the holder

ELIGIBILITY:
Inclusion Criteria:

* • Subject's age ranges from 18-45

  * Having neck discomfort symptoms that were triggered by certain neck positions and by palpating the cervical musculature for at least three months
  * Smartphones addiction >6hours per day

Exclusion Criteria:

* • Pregnancy.

  * Neck pain associated with whiplash injuries or trauma
  * medical red flag history (such as tumour, fracture, metabolic diseases, rheumatoid arthritis and osteoporosis)
  * Neck pain with cervical radiculopathy or neck pain associated with externalized cervical disc herniation.
  * If the patient had previous surgery in the neck area (irrespective of the reason for the operation)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
neck pain intensity | "From enrollment to the end of treatment at 4 weeks"
  using numeric pain rating scale which compose of 11 points from 0 to 10, while zero indicate no pain and 10 indicates maximum unimaginable pain.
pain pressure threshold | "From enrollment to the end of treatment at 4 weeks"
  using algometer

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Outpatient's clinics of the faculty of physical therapy, Benha university, Banhā
  - Faculty of Physical Therapy, Benha University, Banhā